CLINICAL TRIAL: NCT00699309
Title: A Prospective, Non-controlled, Clinical Investigation of the Taperloc® Microplasty™ Hip System
Brief Title: A Clinical Investigation of the Taperloc® Microplasty™ Hip System
Status: Completed | Type: Observational
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: Biomet 13594-115
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Avascular Necrosis
Keywords: Total Hip Replacement; Total Hip Arthroplasty; Minimally Invasive; Microplasty; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Taperloc® Microplasty™ Hip System

SUMMARY:
The purpose of this prospective clinical data-collection is to document the performance and clinical outcomes of the Taperloc® Microplasty™ Hip System.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid arthritis.
* Correction of functional deformity.
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques.
* Revision of previously failed femoral head resurfacing component

Exclusion Criteria:

Absolute contraindications include:

* infection,
* sepsis, and
* osteomyelitis.

Relative contraindications include:

* uncooperative patient or patient with neurologic disorders who are incapable of following directions,
* osteoporosis,
* metabolic disorders which may impair bone formation,
* osteomalacia,
* distant foci of infections which may spread to the implant site,
* rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
* vascular insufficiency, muscular atrophy, or neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring relief from painful or disabling joint disease.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2005-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 5 years

SECONDARY OUTCOMES:
Incidence of revision or removals | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, PhD, Study Director — Director, Clinical Research, Biomet Orthopedics, LLC
Locations (4):
- United States (4):
  - Low Country Bone & Joint Specialists, Beaufort, South Carolina
  - Piedmont Orthopedics, Greenville, South Carolina
  - Texas Center for Joint Replacement, Plano, Texas
  - Arthritis & Sports Orthopaedics, Sterling, Virginia